CLINICAL TRIAL: NCT03175068
Title: Transdiagnostic Brain-Behavior Profiling to Enhance Cognitive Behavioral Therapy Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Heide Klumpp, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-0258; 1R01MH112705-01A1 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder; Social Anxiety Disorder
Keywords: Functional magnetic resonance imaging; Electroencephalography; Cognitive Behavioral Therapy; Supportive Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Phobia, Social | interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (Active Comparator): The clinical psychologist will use a manualized CBT approach tailored to MDD or gSAD. Over a 12-week period sessions will include core CBT strategies -- psychoeducation, cognitive intervention (e.g., cognitive restructuring), behavioral changes (i.e., fear exposure, behavioral activation strategies) and relapse prevention.
  Interventions: Behavioral: CBT
- ST (Placebo Comparator): The clinical psychologist will use an ST approach that resembles client-centered therapy of Carl Rogers (1951) which has been used as a control psychotherapy. The manual is based on supportive psychotherapy principles. Over a 12-week period sessions will emphasize reflective listening and elicitation of affect. In contrast to CBT, therapists allow patients to determine the focus of each session, pulling for emotion, validating emotions when possible, and offering empathetic comments. Therapists will refrain from delineating any CBT theoretical framework and avoided cognitive and behavioral techniques that might overlap with CBT.
  Interventions: Behavioral: ST

INTERVENTIONS:
Behavioral: CBT — CBT works by changing people's attitudes and their behavior by focusing on the thoughts, images, beliefs and attitudes that are held (a person's cognitive processes) and how these processes relate to the way a person behaves, as a way of dealing with emotional problems.
  Other Names: Cognitive Behavioral Therapy
  Arms: CBT
Behavioral: ST — Treatment designed to improve, reinforce, or sustain a patient's physiological well-being or psychological self-esteem and self-reliance
  Other Names: Supportive Therapy
  Arms: ST

SUMMARY:
Many patients with Major Depressive Disorder (MDD) and generalized Social Anxiety Disorder (gSAD) are treated with cognitive behavioral therapy (CBT) but few have meaningful improvement. MDD and gSAD are diseases of brain dysfunction that manifest as impaired emotion regulation; CBT teaches emotion regulation strategies but how it works in the brain remains largely unknown. Individual differences in brain function related to emotion regulation may make some patients better suited for CBT and CBT may remedy the brain dysfunction that underlies these disorders. This project will compare CBT with a placebo psychotherapy (i.e., supportive therapy) in MDD and gSAD to test, validate, and refine brain-based markers and examine mechanisms of change to examine how CBT works and for whom.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) and generalized Social Anxiety Disorder (gSAD) are pervasive major public health problems. These disorders are characterized by emotion dysregulation, an inability or inefficiency to regulate negative and positive affect as reflected in common and disorder-specific symptoms (e.g., attentional bias to negative stimuli, excessive/inappropriate negative thoughts, hyperarousal, anhedonia, emotional blunting). Such dysregulation is believed to result from an imbalance between top-down 'emotion regulating' (ER) frontal nodes central in inhibitory control of bottom-up subcortical 'emotion-generating' (EG) nodes in a Fronto-Limbic Affect Regulation and Emotional Salience (FLARES) network. Therefore, successful treatment would be expected to 'normalize' neurofunctional disturbances in the FLARES network, which can be measured with fMRI and more distal units of brain function -- event-related potentials (ERPs) from electroencephalography, startle potentiation from electromyography (EMG), neurocognitive performance, and use of regulation strategies in daily life via self-report. The overarching objective of the proposed study is to understand how, when, and where CBT works and for whom to tailor treatment to improve clinical outcome.

Without precisely identified "targets" and "predictors" of change, CBT response will continue to be unpredictably varied with few achieving meaningful clinical improvement placing them at risk for relapse and recurrence. Our proposal builds on published data from our lab and others and Preliminary Data which shows FLARES function, as assayed with fMRI, ERPs, EMG, and behaviors, is sensitive to change following CBT.

Importantly, both baseline fMRI and non-fMRI units of brain-behavioral measures predict CBT response better than baseline clinical measures. Such knowledge can lead to more precise interventions aimed at capitalizing on 'strengths' or improving 'deficits' that may each exist before CBT and/or explain why CBT does not work for some patients. The dual development of fMRI ('mechanistic') and non-fMRI ('pragmatic') predictors and indices of therapeutic change is aimed at advancing precision medicine while increasing the clinical utility of 'biomarkers' in the outpatient setting. With this objective, we propose to employ well-validated paradigms to test ER and EG in the context of negative stimuli, reward processes, and fear systems in MDD and gSAD to delineate common and disorder-specific mechanisms of change and predictors of CBT outcome. We will enroll 200 patients: 100 MDD (without comorbid gSAD), 100 gSAD (without comorbid MDD) and randomize them to 12 weeks of manualized CBT or 12 weeks of 'placebo' psychotherapy (supportive therapy) (1:1 ratio). Multiple units of FLARES function will be collected in all patients before (Week 0), during (midway/Week 6) and after treatment (Week 12) to ascertain CBT 'dose' effects, and in 40 healthy controls for comparison. Pre-CBT predictors based on binary (responder/non-responder status) and continuous (extent of change) outcomes will be examined midway (Week 6), immediately after treatment (Week 12), and at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. generally medically and neurologically healthy, including no evidence of mental retardation or serious cognitive impairment that would interfere with protocol adherence and/or task performance
2. between the ages of 18 - 65 years old, inclusive
3. right-handed
4. primary diagnosis of MDD or gSAD based on the SCID DSM-5. Patients will be permitted to have limited comorbid and/or history of internalizing psychopathologies (e.g., generalized anxiety disorder, specific phobia, adjustment disorder)

Exclusion Criteria:

1. personal current or past manic/hypomanic episode or psychotic symptoms
2. active suicidal ideation as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)
3. prior history of standard CBT (failure or success)
4. any current or recent (past 4 weeks) use of medication (prescription or non-prescription) with psychotropic effects
5. psychotherapy other than CBT or psychotropic medication use during the study
6. cognitive dysfunction (traumatic brain injury, mental retardation, dementia)
7. active moderate or severe alcohol and/or substance use disorders

For healthy controls: history or current Axis I disorder.

Additional exclusion criteria for all participants pertaining to the fMRI scan include:

1. presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
2. inability to tolerate small, enclosed spaces without anxiety (e.g., claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
BOLD Effects Measured with Functional Magnetic Resonance Imaging (fMRI) | Weeks 0, 6, and 12
  Patients were randomized to either 12 weeks of cognitive behavioral therapy or supportive therapy. Healthy control (HC) participants did not receive treatment but completed the same assessments at the same time points as patients. Mean BOLD effects in emotion processing and cognitive control tasks at baseline, at mid-point of treatment (for patients)/time interval (for HC), and at end of treatment (for patients)/time interval (for HC). Target areas are analyzed from fMRI scans. The scans were completed on Weeks 0, 6, and 12. Average BOLD effects were calculated for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Heide Klumpp, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Feurer C, Jimmy J, Bhaumik R, Duffecy J, Medrano GR, Ajilore O, Shankman SA, Langenecker SA, Craske MG, Phan KL, Klumpp H. Anterior cingulate cortex activation during attentional control as a transdiagnostic marker of psychotherapy response: a randomized clinical trial. Neuropsychopharmacology. 2022 Jun;47(7):1350-1357. doi: 10.1038/s41386-021-01211-2. Epub 2021 Oct 30. PMID 34718341